CLINICAL TRIAL: NCT01989416
Title: Effectiveness of Chlorhexidine Wipe for Prevention of Multidrug-resistant Organisms in Intensive Care Unit Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Adhiratha Boonyasiri, Doctor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 567-2556-EC4
Record Dates: First submitted 2013-10-13; First posted 2013-11-21 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Antibiotic Resistant Infection
Keywords: colonization
MeSH Terms: interventions — Soaps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soap bathing (Placebo Comparator): ICU patients will be bathing with soap at least once daily
  Interventions: Drug: Soap
- 2% chlorhexidine wipes (Experimental): Use 2% chlorhexidine wipes to clean the patient at least once daily
  Interventions: Drug: 2% chlorhexidine wipe

INTERVENTIONS:
Drug: 2% chlorhexidine wipe — The ICU patients will be bathing with 2% chlorhexidine wipe
  Other Names: chlorhexidine wipe
  Arms: 2% chlorhexidine wipes
Drug: Soap — The ICU patients will be bathing with Soap
  Other Names: Control soap
  Arms: Soap bathing

SUMMARY:
The purpose of this study is to determine 2% chlorhexidine wipes are effective in preventing of colonization of multi-drug resistant bacteria in intensive care unit patients.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the usefulness of bathing with chlorhexidine wipe to reduce the risks of multidrug resistant bacteria acquisition and hospital-acquired bloodstream infection among ICU patients

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Admission in critical care unit eg. ICU, respiratory care unit, Cardiac care unit with in 24 hours
* Expected duration of critical care unit admission > 48 hours

Exclusion Criteria:

* History of chlorhexidine allergy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The overall rate of Multidrug resistant bacteria acquisition at 7 days after received 2% chlorhexidine wipe bathing versus with soap bathing | 7 days after recieved 2% chlorhexidine wipes
  7 days after received 2% chlorhexidine wipes,the microbiology laboratory will process surveillance specimens using either standard culture-based at both nostrils, axillar, groins, rectum

SECONDARY OUTCOMES:
The overall rate of hospital-acquired bloodstream infections per 1000 patient-days with chlorhexidine wipe bathing versus with soap bathing | 48 hours after recieved 2% chlorhexidine wipes

CONTACTS AND LOCATIONS:
Overall Officials: Adhiratha Boonyasiri, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Boonyasiri A, Thaisiam P, Permpikul C, Judaeng T, Suiwongsa B, Apiradeewajeset N, Fakthongphan T, Suddee S, Laoagtipparos W, Thamlikitkul V. Effectiveness of Chlorhexidine Wipes for the Prevention of Multidrug-Resistant Bacterial Colonization and Hospital-Acquired Infections in Intensive Care Unit Patients: A Randomized Trial in Thailand. Infect Control Hosp Epidemiol. 2016 Mar;37(3):245-53. doi: 10.1017/ice.2015.285. PMID 26894621